CLINICAL TRIAL: NCT02947113
Title: Feasibility Trial on Combination of Platinum Doublets and Hypofractionated Radiotherapy for Locally-advanced Stage and / or Inoperable Non-small Cell Lung Carcinoma
Brief Title: Combination of Platinum Doublets and Hypofractionated Radiotherapy in NSCLC
Acronym: HYPOLAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: New studies available with immunotherapy so recruitment is no longer acceptable.
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16HYP; 2016-003790-18 (EudraCT Number); NL57625.031.16 (Other: CCMO)
Record Dates: First submitted 2016-10-14; First posted 2016-10-27 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Cisplatin; Radiation Dose Hypofractionation; Pemetrexed; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy combined with radiotherapy (Experimental): Patients will be treated with two 3-weekly courses of cisplatin (Day 1: 75mg/m2) and pemetrexed (Day 1: 500mg/m2 for non-squamous) or etoposide (Day1-3 100mg/m2 for squamous), together with hypofractionated radiotherapy (24 daily fractions of 2.42 Gy to the involved mediastinal lymph nodes with an integrated boost of 2.75 Gy to the primary tumor).
  Interventions: Drug: Cisplatin; Radiation: hypofractionated radiotherapy; Drug: Pemetrexed; Drug: Etoposide

INTERVENTIONS:
Drug: Cisplatin — Cisplatin will be administrated in a 3-weekly scheme for 2 courses combined with pemetrexed (non-squamous cell lung cancer) or etoposide (squamous cell lung cancer)
Radiation: hypofractionated radiotherapy — Hypofractionated radiotherapy of 24 x 2.75 Gy will be given combined with a 3-weekly scheme of cisplatin and pemetrexed/etoposide
Drug: Pemetrexed — Pemetrexed will be administrated in a combination with cisplatin and hypofractionated radiotherapy (for non-squamous cell lung cancer)
  Other Names: Alimta
Drug: Etoposide — etoposide will be administrated in a combination with cisplatin and hypofractionated radiotherapy (for squamous cell lung cancer)
  Other Names: Etoposin

SUMMARY:
Concurrent chemoradiotherapy is the standard treatment for locally advanced non-small cell lung carcinoma (NSCLC). Different chemotherapy and radiation regimens have been advocated but in general, cisplatin-doublets are deemed standard of care. Decreasing the overall treatment time of irradiation by hypofractionation is thought to increase the efficacy. Extensive experience is available on the combination of daily-dose cisplatin in combination with hypofractionated radiotherapy. However, no data is available on the safety of cisplatin doublets and hypofractionated radiotherapy

DETAILED DESCRIPTION:
Patients presenting with locally advanced NSCLC will be consented to participate in this phase 2 trial that evaluates the concurrent treatment of cisplatin (Day 1: 75mg/m2) and pemetrexed (Day 1: 500mg/m2 for non-squamous cell lung cancer) or etoposide (Day1-3 100mg/m2 for squamous cell lung cancer), 3-weekly regimens, together with radiotherapy (24 daily fractions of 2.42 Gy to the mediastinal lymph nodes with an integrated boost of 2.75 Gy to the primary tumour). An interim analysis is planned following the first cohort of 25 patients to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Male or female aged 18 years or older
* Cytological or histological proven NSCLC stage III or inoperable stage II (cT1-3-3N0-1), according to the 8th edition of the AJCC staging.
* Patients with locoregional recurrent lung tumor following surgery or a second primary cancer are eligible, unless a pneumonectomy was performed.
* Minimum required laboratory data
* Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 5.5 mmol/L.
* Hepatic:

  i. Serum bilirubin ≤ 1.5 times the upper limit of normal (× ULN); alkaline phosphatase (AP), aspartate aminotransferase (ASAT), and alanine aminotransferase (ALAT) ≤ 3.0 × ULN.

ii. This does not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinaemia that is predominantly unconjugated in the absence of evidence of haemolysis or hepatic pathology) who will be allowed in consultation with their physician.

* Renal: GFR ≥ 60 ml/min; if below this threshold a creatinine clearance (CrCL) can be calculated based on the original weight based Cockcroft and Gault formula and should be ≥ 45 ml/min.

Exclusion Criteria:

* WHO performance status ≥ 2
* FEV-1 and DLCO < 35 % of the age- and gender adjusted normal value
* Patients with grade 3 dyspnea or worse at baseline (according to CTCAE version 4.03)
* Prior radiotherapy to the thorax.
* Mean lung dose > 20.0 Gy and/or exceeding other organs-at-risk constraints (page 21).
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of chemotherapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the chemoradiotherapy or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related Adverse events (according to CTCAE v 4.03) | within 3 months FU
  safety defined by the rate of grade 3-5 adverse events

SECONDARY OUTCOMES:
safety defined by the rate of grade 3-4 treatment related adverse events | 3 months
  safety will be assessed by the incidence of grade 3-4 related adverse event (CTCAE v 4.03)
disease control rate | 1 year
progression free survival | 2 years
overall survival | 2 years

OTHER OUTCOMES:
biomarker | through study completion, an average of 2 years
  assessment of circulating cell free tumor DNA for residual disease

CONTACTS AND LOCATIONS:
Overall Officials: Judi van Diessen, MD, Principal Investigator — The Netherlands Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran WJ Jr, Paulus R, Langer CJ, Komaki R, Lee JS, Hauser S, Movsas B, Wasserman T, Rosenthal SA, Gore E, Machtay M, Sause W, Cox JD. Sequential vs. concurrent chemoradiation for stage III non-small cell lung cancer: randomized phase III trial RTOG 9410. J Natl Cancer Inst. 2011 Oct 5;103(19):1452-60. doi: 10.1093/jnci/djr325. Epub 2011 Sep 8. PMID 21903745
- [Background] Kwint M, Uyterlinde W, Nijkamp J, Chen C, de Bois J, Sonke JJ, van den Heuvel M, Knegjens J, van Herk M, Belderbos J. Acute esophagus toxicity in lung cancer patients after intensity modulated radiation therapy and concurrent chemotherapy. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):e223-8. doi: 10.1016/j.ijrobp.2012.03.027. Epub 2012 May 5. PMID 22560551
- [Background] Mauguen A, Le Pechoux C, Saunders MI, Schild SE, Turrisi AT, Baumann M, Sause WT, Ball D, Belani CP, Bonner JA, Zajusz A, Dahlberg SE, Nankivell M, Mandrekar SJ, Paulus R, Behrendt K, Koch R, Bishop JF, Dische S, Arriagada R, De Ruysscher D, Pignon JP. Hyperfractionated or accelerated radiotherapy in lung cancer: an individual patient data meta-analysis. J Clin Oncol. 2012 Aug 1;30(22):2788-97. doi: 10.1200/JCO.2012.41.6677. Epub 2012 Jul 2. PMID 22753901